CLINICAL TRIAL: NCT05631106
Title: Lifestyle Interventions for Vitality and Empowerment in Seniors
Acronym: LIVES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wake Forest University (Other)
Responsible Party: Principal Investigator, Jeff Katula, Professor, Wake Forest University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00024800
Record Dates: First submitted 2022-11-18; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Cognitive Change
MeSH Terms: interventions — Range of Motion, Articular

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stretching, Balance, Range of Motion (Active Comparator): Participants will engage stretching, balance, and range of motion exercises 2 days per week for 12-weeks.
  Interventions: Behavioral: Stretching, Balance, and Range of motion
- High Intensity Interval Resistance Training (Experimental): Participants will perform resistance training exercises at high intensity intervals 2 days per week for 12-weeks.
  Interventions: Behavioral: High Intensity Interval Resistance Training

INTERVENTIONS:
Behavioral: High Intensity Interval Resistance Training — During each group exercise session, the participants will be guided through a 5-minute warm-up, supervised to perform two sets of machine-based leg press, chest press, seated row, and shoulder press exercises at 30% of 1-RM, and guided through a cool-down. Each exercise set will be 40 -seconds in length with instructions to perform as many repetitions as possible followed by a 20-second rest in between sets and a three-minute rest between exercises.
  Arms: High Intensity Interval Resistance Training
Behavioral: Stretching, Balance, and Range of motion — The stretching, balance, and range of motion intervention will include a rotating and varied routine of stretching exercises for large and small muscle groups, and activities to improve balance and range of motion. Participants will attend this intervention twice a week with each session lasting 30 minutes.
  Arms: Stretching, Balance, Range of Motion

SUMMARY:
The goal of this clinical trial is to test a newer type of high intensity interval resistance training in adults 65 years of age or older. The main aims of this study are:

1. To develop study procedures in order to conduct a randomized controlled trial to test the impact of high intensity interval training on cognition in older adults. We will develop procedures for recruitment, screening, data collection, blinded randomization, HIIRT and EA interventions, safety monitoring, and data analyses.
2. To determine the feasibility of using high intensity interval resistance training as an intervention. Feasibility will be shown by; 1) recruiting the target population and meeting our overall patient accrual goal of 30 participants over a 12-week period, 2) achieving an average attendance rate of ≥ 70% of the 24 scheduled sessions in the HIIRT group, 3) at least 80% retention of participants at the final follow-up assessment (week 12), and 4) successful completion of the MRI task (finishing the session with a behavioral accuracy greater than 70%) by at least 80% of participants. Acceptability will be assessed via participants' ratings on a standardized measure of treatment satisfaction and reasons for dropout. Acceptability will be indicated in 2 ways: 70% of the participants report treatment satisfaction on a standard questionnaire, and consistent collection of follow-up data across sites.
3. To examine causal mechanisms and preliminary efficacy. We will examine the relationships among several proposed mediators of the expected treatment effect. We will also examine the mean change and variability of our primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Lives within 20 miles of the school
* Does not plan to travel outside the home geographic area for an extended period during the study participation
* Willing to provide informed consent
* Willing to be randomized to either lifestyle intervention group
* Willing to complete all study procedures and assessments
* No contraindications to exercise
* Capacity to complete physical exercise

Exclusion Criteria:

* Dependent on walking device
* Claustrophobia
* Performs 30 minutes of moderate intensity exercise three times per week for the previous three months
* Joint replacement or orthopedic surgery in the previous 6-months or planning to have surgery in the next 6-months
* Uncontrolled hypertension
* Pathological neurological condition
* Parkinson's disease
* Unstable depression, anxiety, or schizophrenia (medication changes in the past 6 months)
* Experienced a concussion within the last 6 months
* Respiratory disease requiring oxygen
* Cancer requiring treatment
* Osteoarthritis
* Osteopenia or Osteoporosis
* Body mass index under 18
* Muscle wasting disease
* Hypertrophic or dilated cardiomyopathy significant cardiovascular disease (NIHA Class III/IV congestive heart failure, aortic stenosis, history of cardiac arrest, uncontrolled angina)
* Currently receiving physical therapy or cardiopulmonary rehabilitation
* Type I or insulin dependent Type II Diabetes
* Any implanted medical devices that are not compatible with fMRI scans (cardiac pacemaker or implanted cardiac defibrillator (ICD))
* Metal shavings in eyes
* Ferromagnetic piercings that cannot be taken out
* Transdermal patches that cannot be removed
* Cerebral aneurysm clip
* >14 alcoholic drinks in one week
* Not receiving medical clearance after PARQ+
* Evidence of cognitive impairment (Scoring below 32 points on the Telephone Interview of Cognitive Status)
* Site PI/Study Clinician discretion regarding medical status, appropriateness of participation or concern about intervention adherence, clinical judgement

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Executive Functioning | Baseline and 12-weeks
  Executive Functioning will be operationalized as an index of several computer-based tasks assessing aspects of executive functioning: Inhibition (Stroop Test), Updating (The 4-part continuous performance task), and Switching (Shifting attention task, Symbol Digit Coding).
Gradual Continuous Performance Test | Baseline and 12-weeks
  Participants will make continuous responses to target picture stimuli (images of cities among distractor images of mountains). Periodically, a colored border will appear around each location, cuing the participant to attend to either the left or right picture stream. If the currently cued stream differs from their previous focus of attention, the participant will make a saccadic eye movement. At the same time as the color onset, a number will appear at each location. Participants will then make an even/odd discrimination for stimuli appearing at the to-be-attended location.
Functional Magnetic Resonance Imagining | Baseline and 12-weeks
  Participants will complete a 60-minute magnetic resonance imagining session during which will acquire a high-resolution anatomical scan, an echo planar image while participants complete the Gradual Continuous Performance Test. This task is a cognitive task designed to measure the neural correlates of moment-by-moment fluctuations in the efficacy of sustained attention and attention shifting readiness, termed attentional flexibility, a resting state scan, and a diffusion tensor imaging to measure white matter tract integrity.

SECONDARY OUTCOMES:
Brain Derived Neurotrophic Factor | Baseline and 12-weeks
  Blood will be drawn using venipuncture to collect a serum sample. A blood analysis will be performed to examine brain derived neurotrophic factor, a marker suggesting an increase hippocampal neural growth.
The Physical Activity Enjoyment Scale | Baseline and 12-weeks
  The physical activity enjoyment scale captures the extent to which an individual enjoys the physical activities they are currently participating in. The individual is asked to respond to 18 items with bipolar anchors on a 7-point Likert-type scale (e.g., 1=I enjoy it, 7=I hate it; 1=I feel bored, 7=I feel interested).
Community Health Activities Model Program for Seniors Activity Questionnaire for Older Adults | Baseline and 12-weeks
  This physical activity questionnaire tasks participants with reporting the extent to which they participated in various occupational, transport, leisure time, and home physical activities in the previous 4 weeks (e.g., "In a typical or normal week during the past 4 weeks, did you do heavy gardening?"). If the participant indicates "yes" they next indicate the weekly frequency and duration of the activity. Following scoring, the scale produces variables capturing average weekly frequency, duration, and caloric expenditure for both total physical activity and exercise-specific activities.
Basic Psychological Need Satisfaction and Frustration Scales | Baseline and 12-weeks
  he BPNSFS reflect the extent to which an individual experiences satisfaction and frustration in achieving the core human needs of relatedness, competence, and autonomy. Participants respond to 24 questions (e.g., "I feel a sense of choice and freedom in the things I undertake") on a 5-point Likert-type scale where 1 indicates "Not True at All" and 5 indicates "Completely True". The scale produces 6 subscale scores, including both frustration and satisfaction subscales for autonomy, competence, and satisfaction. Each subscale is computed as the sum of four questionnaire items, with scores ranging from 4-20, with higher scores reflecting greater satisfaction or frustration.
SF-36 Health Questionnaire | Baseline and 12-weeks
  The SF-36 is a generic measure of health status/health-related quality of life that consists of two norm-based composite T-scales, mental health and physical function, and 8 subscales: physical functioning, mental health, role-physical, role-emotional, bodily pain, general health, vitality, and social functioning.
400 Meter Walk Test | Baseline and 12-weeks
  The 400 meter walk test assesses walking speed and endurance in older adults on a 20 meter course. The timed walk covers 10 laps totaling 400 meters.
Short Physical Performance Battery | Baseline and 12-weeks
  This measure assesses lower extremity functioning.
Stroop Test | Baseline and 12-weeks
  This is a three part test. Participants will be asked to respond the words "RED", "GREEN", "YELLOW", "BLUE", and "GREEN" in different colors according to the instructions provided for each part.
Symbol Digit Coding | Baseline and 12-weeks
  The symbol digit coding test measures complex information processing accuracy, complex attention, visual-perceptual speed, and information processing speed.
Four-Part Continuous Performance Test | Baseline and 12-weeks
  The four-part continuous performance is a test that measures the participant's working memory and sustained attention.
Shifting Attention Test | Baseline and 12-weeks
  The shifting attention test is a measure of ability to shift from one instruction set to another quickly and accurately. Participants will be instructed to match geometric objects either by shape or by color.

IPD SHARING:
Plan to Share IPD: No